CLINICAL TRIAL: NCT03306810
Title: Recognition and Treatment of Dysglycemia in Elective Knee and Hip Arthroplasties. AGS - Acute Glucose Service
Brief Title: Recognition and Treatment of Dysglycemia. AGS - Acute Glucose Service
Acronym: AGS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Responsible Party: Principal Investigator, Marjo Soini, CRA, Joint Authority for Päijät-Häme Social and Health Care
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Q321dnro 47/17
Record Dates: First submitted 2017-09-19; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Dysglycemia; Arthroplasty Complications
Keywords: Perioperative complications; Dysglycemia management team; Nurse Practitioner; Hospital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AG service (Active Comparator): In the "Active Comparator Arm": Screening, follow-up and treatment of dysglycemias in the elective orthopedic prosthetic surgery (knee / hip) patients in the Päijät-Häme Central hospital will be optimized and individualized in the patients in personal manner.
  Interventions: Other: AG service
- Without AG service (No Intervention): In the "No intervention Arm": Screening, follow-up and treatment of dysglycemias in the elective orthopedic prosthetic surgery (knee / hip) patients follows the current protocol of Päijät-Häme Central hospital.

INTERVENTIONS:
Other: AG service — The AG service group is divided to two 200 patients groups: 1) with AGS 2) with AGS extended to first control in 3 months (AG- nurse may be contacted by phone). Patients are followed up up to 5 years.
  Arms: AG service

SUMMARY:
AGS (Acute Glucose Service ) is an inpatient glucose management service consisting of Nurse Practitioner and physician. Team manages not - consulted- based preoperative assessment, perioperative glucose control, patient education and supervision, but also transition of care postoperatively. The goal is to detect and treat dysglycemias , but also provide an active and constantly ongoing education to other hospital teams.

AGS improves better overall- survival of arthroplastic patients and is an effective way to recognize and treat dysglycemias and to organize constantly ongoing education.

DETAILED DESCRIPTION:
600 elective knee and hip arthroplastic patients are collected. 200 patients before AG- service will be compared to 400 patients after AGS. The latter group is divided to two 200 patients groups: 1) with AGS 2) with AGS extended to first control in 3 months (AG- nurse may be contacted by phone). Patients are followed up up to 5 years. Controls will be held after 3 months, 1 year and 5 years after operation including B-Hba1c, 15 D Quality of life assessment and patient interview.

There are several aims of the team and study: to detect, diagnose and optimize treatment (including medication) of diabetic/ dysglycemic patients from preoperative assessment 1 week before operation to postoperative care. With blood glucose target 42 - 86 mmol/mol results better overall survival, lesser complications (i.e. infections, cardiovascular or renal complications) and shorter length of hospital stay. Other aim is to find undiagnosed diabetics or those at risk of developing diabetes. One aim is to find risk factors, which lead to stress hyperglycemia during perioperative period or diabetes in 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years
* Elective knee and hip arthroplasty patients

Exclusion Criteria:

* Patients who are incompetent to give informed consent
* Patients who are incompetent to assess their Quality-of-Life personally

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 1-5 years
  Improved survival

SECONDARY OUTCOMES:
Complications | 1-5 years
  Less complications after AG-service

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Ylikoski, MD, Principal Investigator — Päijät Häme Central Hospital
Locations (1):
- Päijät-Häme Central Hospital, Lahti, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ylikoski M, Jokinen JJ, Lahtela J, Kauppi MJ, Huhtala H, Immonen H, Tiihonen R. Perioperative hyperglycaemia in elective arthroplasties. Should we do better? Acta Anaesthesiol Scand. 2020 Oct;64(9):1253-1261. doi: 10.1111/aas.13666. Epub 2020 Jul 30. PMID 32615649